CLINICAL TRIAL: NCT03790657
Title: Cerebral Networks of Locomotor Learning and Retention in Older Adults
Brief Title: CONTROL Walking Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3115-R; I01RX003115 (NIH)
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: aging; walking; brain; electrical stimulation

STUDY DESIGN:
Intervention Model Description: Participants will randomized to one of two dosages of transcranial direct current stimulation (tDCS): Dosage A or Dosage B
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told which dosage group they are assigned to. Outcomes Assessors will not be told which dosage group the participant was randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): 20 minutes of mild electrical stimulation delivered to the frontal region of the brain during practice of a complex walking task
  Interventions: Behavioral: practice of a complex walking task; Device: Active transcranial direct current stimulation (Active tDCS)
- Sham tDCS (Sham Comparator): 30 seconds of mild electrical stimulation delivered to the frontal region of the brain during practice of a complex walking task
  Interventions: Behavioral: practice of a complex walking task; Device: Sham transcranial direct current stimulation (Sham tDCS)

INTERVENTIONS:
Behavioral: practice of a complex walking task — walking over obstacles
Device: Active transcranial direct current stimulation (Active tDCS) — mild electrical stimulation delivered to the frontal region of the brain
  Arms: Active tDCS
Device: Sham transcranial direct current stimulation (Sham tDCS) — 30 seconds of mild electrical stimulation delivered to the frontal region of the brain
  Arms: Sham tDCS

SUMMARY:
Older adults often experience substantial deficits in walking ability, especially for walking tasks that are more complex such as obstacle crossing. This is due in part to changes in the brain that make performance of physical and cognitive tasks more difficult. Rehabilitation can help to improve walking ability, but effective rehabilitation is time consuming and expensive. New approaches are needed to improve the efficiency of rehabilitation so that gains in walking ability are widely attainable. A promising strategy is to focus on enhancing motor learning, which is defined as improved ability to perform a motor task due to practice or experience. The investigators will investigate the use of non-invasive brain stimulation to increase motor learning and retention of the newly learned walking skills. The investigators will also use neuroimaging to assess brain characteristics that explain how motor learning works. The knowledge gained from this study is expected to contribute to better understanding of mechanistic targets and intervention approaches to improve rehabilitation of walking.

DETAILED DESCRIPTION:
Aging often leads to substantial declines in walking function, especially for walking tasks that are more complex such as obstacle crossing. This is due in part to a lack of continued practice of complex walking (sedentary lifestyle) combined with age-related deficits of brain structure and the integrity of brain networks. Neurorehabilitation can contribute to recovery of lost walking function in older adults, but major and persistent improvements are elusive. A cornerstone of neurorehabilitation is motor learning, defined as an enduring change in the ability to perform a motor task due to practice or experience. Unfortunately, in most clinical settings, the time and cost demands of delivering a sufficiently intensive motor learning intervention is not feasible. There is a need for research to develop strategies for enhancing motor learning of walking ("locomotor learning") in order to improve the effectiveness of neurorehabilitation.

The objective of this study is to use non-invasive brain stimulation to augment locomotor learning and to investigate brain networks that are responsible for locomotor learning in mobility-compromised older adults. The investigators have shown that frontal brain regions, particularly prefrontal cortex, are crucial to control of complex walking tasks. The investigators' neuroimaging and neuromodulation studies also show that prefrontal cortex structure and network connectivity are important for acquisition and consolidation of new motor skills. However, a major gap exists regarding learning of walking tasks. The proposed study is designed to address this gap. The investigators' pilot data from older adults shows that prefrontal transcranial direct current stimulation (tDCS) administered during learning of a complex obstacle walking task contributes to multi-day retention of task performance. In the proposed study the investigators will build upon this pilot work by conducting a full scale trial that also investigates mechanisms related to brain structure, functional activity, and network connectivity. The investigators will address the following specific aims:

Specific Aim 1: Determine the extent to which prefrontal tDCS augments the effect of task practice for retention of performance on a complex obstacle walking task.

Specific Aim 2: Determine the extent to which retention of performance is associated with individual differences in baseline and practice-induced changes in brain measures (including gray matter volume and brain network segregation).

Specific Aim 3: Investigate the extent to which tDCS modifies resting state network segregation.

The investigators anticipate that prefrontal tDCS will augment retention of locomotor learning, and that the data will provide the first evidence of specific brain mechanisms responsible for locomotor learning/retention in older adults with mobility deficits. This new knowledge will provide a clinically feasible intervention approach as well as reveal mechanistic targets for future interventions to enhance locomotor learning and retention.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* preferred 10m walking speed < 1.1 m/s
* self-report of "some difficulty with walking tasks, such as becoming tired when walking a quarter mile, or when climbing two flights of stairs, or when performing household chores."
* Willingness to be randomized to either study group and to participate in all aspects of study assessment and intervention

Exclusion Criteria:

* Diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition (Alzheimer's, Parkinson's, stroke, etc.)
* Contraindications to non-invasive brain stimulation (e.g., metal in head, wound on scalp)
* Contraindications to magnetic resonance imaging (e.g., metal in body, claustrophobia, etc).
* Use of medications affecting the central nervous system
* severe arthritis, such as awaiting joint replacement
* severe obesity (body mass index > 35)
* current cardiovascular, lung or renal disease; diabetes; terminal illness
* myocardial infarction or major heart surgery in the previous year
* cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis (e.g., early stage breast or prostate cancer)
* current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* bone fracture or joint replacement in the previous six months
* current participation in physical therapy for lower extremity function or cardiopulmonary rehabilitation
* current enrollment in any clinical trial
* difficulty communicating with study personnel, and/or non-English speaking
* planning to relocate out of the area during the study period
* clinical judgment of investigative team regarding safety or non-compliance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Clark, DSc, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset will be created and shared pursuant to a Data Use Agreement appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The Limited Dataset will be completed after the study is completed and primary/secondary data accepted for publication.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened to ensure they met all inclusion/exclusion criteria, did not have major disease or injury affecting brain function or walking function, were medically stable, and could safely participate in the study protocol.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 34 | 38
Completed | 32 | 36
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: These numbers are those who passed the onsite screening visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: These numbers are those who passed the onsite screening visit.
  years | 72.97 (5.65) | 75.83 (8.06) | 74.49 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: These numbers are those who passed the onsite screening visit.
  Participants
    Female | 8 | 17 | 25
    Male | 24 | 19 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: These numbers are those who passed the onsite screening visit.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 30 | 33 | 63
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: These numbers are those who passed the onsite screening visit.
  Participants
    Hispanic or Latino | 2 | 2 | 4
    Not Hispanic or Latino | 30 | 34 | 64
    Unknown or Not Reported | 0 | 0 | 0
Walking speed [Mean (Standard Deviation); unit: meters per second] — preferred walking speed over 10 meters Population: These numbers are those who passed the onsite screening visit.
  meters per second | 1.25 (0.23) | 1.19 (0.19) | 1.22 (0.21)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The scores range between 0 to 30 points; higher values represent a better outcome. Population: These numbers are those who passed the onsite screening visit.
  units on a scale | 26.41 (1.88) | 26.58 (2.6) | 26.5 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed Change From Baseline
Description: Change in the fastest safe walking speed over a complex walking course
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 32 | 36
meters per second | 0.033 (0.097) | 0.041 (0.104)

2. Secondary Outcome: Prefrontal Cortex Gray Matter Volume Change From Baseline
Description: Change in the volume of gray matter in the prefrontal cortex, as measured by MRI
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Population: Some participants did not complete the MRI assessment at baseline or at follow-up due to technical or logistical difficulties.
Measure: Mean (Standard Deviation); unit: cubic millimeters
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 31 | 32
cubic millimeters | -14.66 (81.75) | -3.45 (90.60)

3. Secondary Outcome: Brain Resting State Network Segregation (Z-transformed Correlation Coefficient)
Description: Resting-state functional MRI was used to measure the segregation of large-scale brain networks. Connectivity strength was quantified using Fisher z-transformed correlation coefficients, averaged across regions of interest within each network. Results are reported as mean z-scores for each group. Higher values reflect greater segregation (i.e., stronger within-network compared to between-network connectivity).
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Population: A total of 65 participants underwent MRI imaging, of which only 50 participants were included. Eight participants were missing either baseline or post-assessment scan. Four participants did not complete all necessary scanning sequences.
Measure: Mean (Standard Deviation); unit: z-transformed correlation coefficient
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 25 | 25
z-transformed correlation coefficient | -.0017 (.0253) | -.0002 (.0215)

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 8 weeks
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/36
Other Adverse Events (participants affected / at risk) | 1/32 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS (N=32) | Sham tDCS (N=36)
Musculoskeletal injury (not serious) (Musculoskeletal and connective tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03790657/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03790657/ICF_000.pdf